CLINICAL TRIAL: NCT03823482
Title: Effect of Regional Anesthesia With Lidocaine on Perioperative Levels of Interleukin-1β, Interleukin-6 and Tumor Necrosis Factor-α in Blood and Cerebrospinal Fluid in Cerebral Aneurysm Patients
Brief Title: Lidocaine and Perioperative Cytokine Levels in Blood and Cerebrospinal Fluid in Cerebral Aneurysm Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Marijana Matas, Principal Investigator, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 51
Record Dates: First submitted 2019-01-24; First posted 2019-01-30 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Aneurysm, Cerebral
Keywords: aneurysm, cerebral; inflammation mediators; lidocaine, hydrochloride
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Lidocaine; Anesthesia, Conduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): Participants in lidocaine group, following induction to general anesthesia, will have lidocaine 2% 4 mg/kg administered as regional anesthesia of the scalp prior to Mayfield frame placement and lidocaine 1% 40 mg topically to the throat prior to direct laryngoscopy and endotracheal intubation. Maximum dosage of lidocaine won't exceed 400 mg.
  Interventions: Drug: Lidocaine
- Control group (No Intervention): Participants in control group will have general anesthesia without lidocaine administration.

INTERVENTIONS:
Drug: Lidocaine — Administration of lidocaine 2% 4 mg/kg administered as regional anesthesia of the scalp prior to Mayfield frame placement and lidocaine 1% 40 mg topically to the throat prior to direct laryngoscopy and endotracheal intubation.
  Other Names: Regional anesthesia
  Arms: Lidocaine group

SUMMARY:
Cerebral aneurysm surgery has significant mortality and morbidity rate. Inflammation plays a key role in the pathogenesis of intracranial aneurysms, their rupture, subarachnoid haemorrhage and neurologic complications. Brain injury activates immune cells and triggers cytokine release. Cytokine level in blood and cerebrospinal fluid is an indicator of inflammatory response. Cytokines contribute to secondary brain injury and can worsen the outcome of the treatment. Preventing secondary brain injury by modulating inflammatory response represents a therapeutic target. Lidocaine is local anesthetic that can be used in neurosurgery for regional anesthesia of the scalp and for topical anesthesia of the throat prior to direct laryngoscopy and endotracheal intubation. Except analgetic, lidocaine has systemic anti-inflammatory and neuroprotective effect. It acts through several mechanisms on various types of immune cells producing immunosuppressing effect. Lidocaine can act on activated microglia within central nervous system causing attenuation of immune response.

Primary aim of this prospective randomized trial is to determine influence of lidocaine administration on inflammatory cytokine levels in serum and cerebrospinal fluid during and following cerebral aneurysm surgery. Secondary aim is to determine possible correlation between levels of cytokines and incidence of neurologic and infectious postoperative complications. For that purpose, postoperative neurological clinical status will be recorded. Signs of vasospasm and pathological postoperative brain CT scan findings will be recorded. Incidence of meningitis, pneumonia and sepsis in postoperative period will also be analyzed.

Hypothesis of this trial is that lidocaine administration during cerebral aneurysm surgery would significantly change levels of pro-inflammatory cytokines in cerebrospinal fluid and serum. Lower concentrations of pro-inflammatory cytokines can possibly contribute to better outcome and significantly lower incidence of postoperative complications. Enzyme-immunochemical analysis will be used to measure levels of interleukin-1β, interleukin-6 and tumor necrosis factor-α in cerebrospinal fluid and serum. Investigation group will have, during cerebrovascular surgery under general anesthesia, regional anesthesia of the scalp and topical anesthesia of the throat prior to laryngoscopy, all done with lidocaine. Control group will have general anesthesia without lidocaine administration.

ELIGIBILITY:
Inclusion Criteria:

* ASA ( American Society of Anesthesiologists) grading status I-III,
* scheduled for cerebral aneurysm surgery under general anesthesia,
* signed informed consent for participating in the research.

Exclusion Criteria:

* poorly controlled chronic or acute cardiovascular, respiratory or autoimmune disease,
* acute infectious disease,
* renal or hepatic insufficiency,
* preoperative Glasgow Coma Scale score lower than 15,
* allergic reaction to any of the medications in protocol,
* pregnancy
* refusal to participate in the research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in concentrations of interleukin-1β | Up to 24 hours after anesthesia induction.
  Concentrations of IL-1β in pg/ml in cerebrospinal fluid and serum measured by enzyme-linked immunosorbent assay
Change in concentrations of interleukin-6 | Up to 24 hours after anesthesia induction.
  Concentrations of IL-6 in pg/ml in cerebrospinal fluid and serum measured by enzyme-linked immunosorbent assay
Change in concentrations of tumor necrosis factor α | Up to 24 hours after anesthesia induction.
  Concentrations of TNF-α in pg/ml in cerebrospinal fluid and serum measured by enzyme-linked immunosorbent assay

SECONDARY OUTCOMES:
Incidence of new motoric deficit | Up to one week postoperatively
  Clinical assessment of neurologic status incidence of generalized epileptic seizure, incidence of vasospasm, pathological finding on brain computerized tomography ( ischemia, edema, bleeding, hydrocephalus).
Incidence of generalized epileptic seizure | Up to one week postoperatively
  Clinical assessment to diagnose generalized epileptic seizure
Incidence of vasospasm | Up to one week postoperatively
  Flow velocity over middle cerebral artery more than 180 cm/s measured by transcranial ultrasound
Incidence of pathological computerized tomography brain scan | Up to one week postoperatively
  Findings of edema, ischemia, bleeding or hydrocephalus on brain CT scan

OTHER OUTCOMES:
Incidence of meningitis, pneumonia and sepsis | Up to one week postoperatively
  Clinical signs and laboratory findings for diagnosing infectious complications

CONTACTS AND LOCATIONS:
Locations (1):
- UHCZagreb, Zagreb, Croatia

REFERENCES:
- [Background] Chaki T, Sugino S, Janicki PK, Ishioka Y, Hatakeyama Y, Hayase T, Kaneuchi-Yamashita M, Kohri N, Yamakage M. Efficacy and Safety of a Lidocaine and Ropivacaine Mixture for Scalp Nerve Block and Local Infiltration Anesthesia in Patients Undergoing Awake Craniotomy. J Neurosurg Anesthesiol. 2016 Jan;28(1):1-5. doi: 10.1097/ANA.0000000000000149. PMID 25493926
- [Background] Guilfoyle MR, Helmy A, Duane D, Hutchinson PJA. Regional scalp block for postcraniotomy analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 May;116(5):1093-1102. doi: 10.1213/ANE.0b013e3182863c22. Epub 2013 Mar 11. PMID 23477962
- [Background] Leng T, Gao X, Dilger JP, Lin J. Neuroprotective effect of lidocaine: is there clinical potential? Int J Physiol Pathophysiol Pharmacol. 2016 Apr 25;8(1):9-13. eCollection 2016. PMID 27186318
- [Background] Hollmann MW, Durieux ME. Local anesthetics and the inflammatory response: a new therapeutic indication? Anesthesiology. 2000 Sep;93(3):858-75. doi: 10.1097/00000542-200009000-00038. No abstract available. PMID 10969322
- [Background] Jeong HJ, Lin D, Li L, Zuo Z. Delayed treatment with lidocaine reduces mouse microglial cell injury and cytokine production after stimulation with lipopolysaccharide and interferon gamma. Anesth Analg. 2012 Apr;114(4):856-61. doi: 10.1213/ANE.0b013e3182460ab5. Epub 2012 Jan 16. PMID 22253275
- [Background] Pawlowska E, Szczepanska J, Wisniewski K, Tokarz P, Jaskolski DJ, Blasiak J. NF-kappaB-Mediated Inflammation in the Pathogenesis of Intracranial Aneurysm and Subarachnoid Hemorrhage. Does Autophagy Play a Role? Int J Mol Sci. 2018 Apr 19;19(4):1245. doi: 10.3390/ijms19041245. PMID 29671828
- [Background] Aoki T, Nishimura M. Targeting chronic inflammation in cerebral aneurysms: focusing on NF-kappaB as a putative target of medical therapy. Expert Opin Ther Targets. 2010 Mar;14(3):265-73. doi: 10.1517/14728221003586836. PMID 20128708
- [Background] Mutlu LK, Woiciechowsky C, Bechmann I. Inflammatory response after neurosurgery. Best Pract Res Clin Anaesthesiol. 2004 Sep;18(3):407-24. doi: 10.1016/j.bpa.2003.12.003. PMID 15212336
- [Background] Chaudhry SR, Stoffel-Wagner B, Kinfe TM, Guresir E, Vatter H, Dietrich D, Lamprecht A, Muhammad S. Elevated Systemic IL-6 Levels in Patients with Aneurysmal Subarachnoid Hemorrhage Is an Unspecific Marker for Post-SAH Complications. Int J Mol Sci. 2017 Dec 1;18(12):2580. doi: 10.3390/ijms18122580. PMID 29194369
- [Background] Osborn I, Sebeo J. "Scalp block" during craniotomy: a classic technique revisited. J Neurosurg Anesthesiol. 2010 Jul;22(3):187-94. doi: 10.1097/ANA.0b013e3181d48846. PMID 20479675
- [Background] Hopkins SJ, McMahon CJ, Singh N, Galea J, Hoadley M, Scarth S, Patel H, Vail A, Hulme S, Rothwell NJ, King AT, Tyrrell PJ. Cerebrospinal fluid and plasma cytokines after subarachnoid haemorrhage: CSF interleukin-6 may be an early marker of infection. J Neuroinflammation. 2012 Nov 23;9:255. doi: 10.1186/1742-2094-9-255. PMID 23176037
- [Derived] Matas M, Sotosek V, Kozmar A, Likic R, Sekulic A. Effect of local anesthesia with lidocaine on perioperative proinflammatory cytokine levels in plasma and cerebrospinal fluid in cerebral aneurysm patients: Study protocol for a randomized clinical trial. Medicine (Baltimore). 2019 Oct;98(42):e17450. doi: 10.1097/MD.0000000000017450. PMID 31626100